CLINICAL TRIAL: NCT02643043
Title: UC-GENOME: Urothelial Cancer-GENOmic Analysis to iMprove Patient Outcomes and rEsearch: Hoosier Cancer Research Network GU15-217
Brief Title: UC-GENOME: Urothelial Cancer-GENOmic Analysis to iMprove Patient Outcomes and rEsearch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Milowsky, MD (Other)
Collaborators: Bladder Cancer Advocacy Network (Other); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Matthew Milowsky, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HCRN GU15-217
Record Dates: First submitted 2015-12-18; First posted 2015-12-30 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Urethral Cancer; Cancer of the Ureter
Keywords: Next Generation Sequencing; Genomic Analysis
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC Subjects (Other): Subjects with confirmed metastatic urothelial cancer willing to participate in biospecimen collection (tissue and blood) for genetic studies.
  Interventions: Other: Biospecimen Collection

INTERVENTIONS:
Other: Biospecimen Collection — Subjects consent to provide access to archival tumor tissue and whole blood samples for genetic analysis. Subjects also consent to the indefinite use of their specimens and linked clinical information for ongoing or future research related to metastatic urothelial cancer.

SUMMARY:
This comprehensive genomic analysis and biospecimen repository study incorporates Next Generation Sequencing (NGS) of archival tumor tissue from 200 subjects with metastatic urothelial cancer in support of several parallel goals. The immediate goal involves generation of a comprehensive report identifying subject specific genetic mutations and/or alterations based on NGS. Additionally, DNA and RNA extracted from tumor specimens and any remaining blocks/slides from the NGS will be stored for future research. Long-term, the goal of this endeavor is to support collaborative translational research projects in metastatic urothelial cancer by allowing investigators to interrogate abstracted coded clinical data linked to data from any biospecimen studies.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

STUDY PLAN:

SUBJECT IDENTIFICATION AND CONSENT:

Sites may approach all subjects who attend an appointment for evaluation of metastatic urothelial cancer for inclusion. Study staff review consent documents with potential subjects and answer any and all questions. If a subject desires additional time or wishes to delay enrollment in the study, he/she is given a copy of the consent document and informed about how to ask questions or enroll at a later date. If the subject chooses to participate in the study, he or she signs the consent, and is given a copy for his or her own records.

BIOSPECIMEN COLLECTION AND PROCESSING:

When subjects are consented for entry into this study, they consent to access of any archival tumor tissue (whether from the primary or any metastatic site) for genetic analysis. This tissue is not de-identified at the time of testing so that a subject specific report may be generated and sent to the treating physician. Further, subjects consent to the indefinite use of their specimens and linked clinical information for ongoing or future biomedical research. Additionally, sites inform subjects during the consent process that researchers may use their information for genetic research including research on somatic or germline mutations. The specimens and report provided to HCRN are de-identified and future analyses will be performed on coded (de-identified) data/specimens.

Collection of Archived Tumor Samples:

* After the subject is consented, sites will request primary and/or metastatic archived tumor tissue. The tissue specimen sent may come in the form of a block or slides. Needle biopsy is also acceptable.
* Each institution can use its own standard operating procedure for the preparation of the FFPE material. Each participating site will ship specimens accessed under GU15-217 directly to the lab performing the NGS analysis. Sites will also request corresponding pathology report(s). A de-identified pathology report will then be sent to HCRN with the tissue.

Collection of Blood for Research Purposes Only:

* Each subject will have 47 mL of blood collected and banked for future testing. 10mL of the sample will be used for plasma for banking. 17 mL of the sample will be used for PBMC isolation and cryopreservation. 20mL of the sample will be used for plasma for cfDNA. Any DNA analysis of blood (including possible germline analysis) is for research purposes only and will be performed on coded (de-identified) samples.

Report Generation:

* The subject specific report generated includes a summary of genomic alterations highlighting those variations considered potentially actionable, a concise discussion of the molecular analyses, a list of potential clinical trials incorporating relevant targeted agents, and potential therapeutic options based on the specific alterations discovered along with associated levels of evidence for each. The selection of clinical trials and levels of evidence provided are based on extensive review and analysis of the literature as well as a BCGC convened panel of experts in bladder cancer. This BCGC expert panel will work with the NGS lab to ensure that all potential clinical trials are represented in the individual subject reports.

Storage for Future Research:

* The BCAN Biobank at Hoosier Cancer Research Network (HCRN) will store DNA and RNA isolated for the study, additional FFPE and any biospecimens remaining after the NGS. If at any point a subject wishes to withdraw from the study, the subject will contact their study physician. HCRN will destroy any specimens that it may link to the subject. Once specimens have been stripped of all identifying information or links to identifying information they cannot be recalled to be destroyed.

COMMUNICATION OF NGS RESULTS TO PROVIDER AND SUBJECT:

After NGS testing is complete, a subject specific report will be provided to the subject's treating physician either in hard copy and/or via on-line portal (typically within 14 business days from receipt of tumor tissue) and a de-identified report to HCRN. If an addendum is made to a report, an updated report will be provided to the treating physician and HCRN in the manner described above. During the informed consent process, sites inform each subject that his or her physician will communicate results of the genetic testing on their tumor specimens. Along with the results that are communicated, the subjects' treating physician will explain the implications of their testing results, including whether their genetic profiles render them potentially eligible for a specific therapy or clinical trial.

Sites also inform subjects that researchers will store any specimens remaining after genetic profiling of their tumor is complete. Storage continues indefinitely for future biomedical research. This may include development of commercial products from their specimens.

Sites must explain to subjects that although a blood sample is being obtained, this study is not aimed at discovering germline mutations. Sites must emphasize that genetic analyses performed within this study should not be construed as genetic testing for genetic mutations associated with hereditary cancer susceptibility. Nevertheless, because NGS may be performed on blood, it is possible that a germline mutation that predisposes a subject to cancer will incidentally be discovered. Subjects will not receive any information about such mutations, however, as this analysis will be performed on de-identified samples.

ABSTRACTION OF MEDICAL RECORDS:

Research staff at each site abstracts clinical information from each subject and enters the information into the web based clinical research platform (EDC system). Data abstracted includes details on the following: demographics, cancer diagnosis, cancer stage, surgical and medical management, any treatment decisions made in response to the NGS results communicated to the physician and any response/longer term outcome data as a result of these treatment decisions.

ACCESS TO DATA/SPECIMENS FOR FUTURE RESEARCH:

The database links coded clinical and genetic data, creating a biospecimen and data repository. These data, along with biospecimens stored at HCRN, will ultimately be available for researchers with BCGC-approved and IRB-approved studies allowing access to these data/specimens, and with HCRN managing the data, protecting the confidentiality of study subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following applicable inclusion criteria to participate in this study:

* IRB-approved written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization for release of personal health information; NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Histologically or cytologically confirmed urothelial cancer of the bladder, urethra, ureter, or renal pelvis.
* Metastatic urothelial cancer as defined by M1 (distant metastatic disease) and/or N3 (nodes outside of the true pelvis) at the time of registration.
* Tumor tissue available and suitable for molecular analyses from at least one of the following sources:

  * Tissue previously stored at enrolling institution
  * Tissue previously stored at an outside institution (other than enrolling institution)
* The tissue specimen may come in the form of a block or slides accessed under UC-GENOME from enrolled subjects. Needle biopsy is also acceptable. Details regarding collection requirements, processing and shipping can be found in the Correlative Laboratory Manual (CLM).
* Willing to provide access to tissue and blood for future research, including genetic studies.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Unwilling or unable to provide informed consent.
* Affected by dementia, altered mental status, or any psychiatric or co-morbid condition that would prohibit the understanding or rendering of informed consent, as determined by treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who receive NGS and have a personalized report generated with potential treatment options | From date of consent to receipt of NGS report (estimate 14 days)
  Subject-specific report that includes a summary of genomic alterations and potential therapeutic options based on the specific alterations and evidence discovered.
Collection of tissue and blood samples from subjects receiving treatment for urothelial cancer | From date of consent and retained indefinitely (estimate 10 years)
  Tissue and blood samples will be preserved and stored in a biorepository that cancer investigators can access for future IRB approved translational studies

SECONDARY OUTCOMES:
Proportion of subjects whose personalized NGS report includes targeted therapy treatment options | From date of consent to receipt of NGS report by treating physician (estimate 14 days)
  Subjects whose treatment options include targeted therapy, of either approved or investigational drugs
Proportion of subjects whose personalized NGS report includes potential clinical trial options | From date of consent to receipt of NGS report by treating physician (estimate 14 days)
  Subjects who enroll in a clinical trial based on NGS results.
Proportion of subjects who receive targeted therapy | From date of consent to receipt of NGS report by treating physician (estimate 14 days)
  Subjects who receive targeted therapy, outside of a clinical trial, based on NGS results
Collect comprehensive demographic data for all subjects enrolled in this clinical trial | From date of consent until end of therapy (assessed up to 2 years)
  Subject demographic characteristics compiled and recorded in a data repository, maintained in a secure platform, that will provide an archive for future research.
Collect comprehensive treatment histories for all subjects enrolled in this clinical trial | From date of consent until end of therapy (assessed up to 2 years)
  Subject treatment histories compiled and recorded in a data repository, maintained in a secure platform, that will provide an archive for future research.
Collect comprehensive clinical outcomes for all subjects enrolled in this clinical trial | From date of consent until end of therapy (assessed up to 2 years)
  Subject clinical outcomes data compiled and recorded in a data repository, maintained in a secure platform, that will provide an archive for future research.
Research projects resulting from biospecimen and data repository | From study close until all biospecimens and data have been utilized (estimate 10 years)
  Number and type of clinical trials and basic/translational science or other research projects initiated, based on the biospecimen and data repository
Overall Survival (OS) | From treatment initiation until death as a result of any cause, up to 60 months
  Compare the overall survival for patients with metastatic urothelial cancer who received a treatment based on the NGS results (on or off of a clinical trial) to those patients who did not

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Milowsky, M.D., Study Chair — Hoosier Cancer Research Network
Locations (8):
- United States (8):
  - University of Southern Cailfornia, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Washignton/Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org